CLINICAL TRIAL: NCT02412943
Title: PAPP-A2 Enzyme Replacement Therapy Using Plasma Transfusion
Brief Title: Pappalysin 2 (PAPP-A2) Enzyme Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PAPPA2 Replacement
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Short Stature, Idiopathic
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PAPP-A2 Enzyme Replacement (Experimental): A 20 cc/kg transfusion of Fresh Frozen Plasma will be given over 3 hours on day 0.
  Interventions: Other: Fresh Frozen Plasma

INTERVENTIONS:
Other: Fresh Frozen Plasma — Liquid portion of human blood that was centrifuged, separated, and frozen solid within 6 hours of collection

SUMMARY:
This study evaluates the transfusion of fresh frozen plasma containing the enzyme PAPP-A2 into the a female adult. This female adult has a mutated version of PAPP-A2 that prevents the unbinding of IGF-1 from IGF binding proteins. The investigator's hypothesize that transfusion of plasma with donor PAPP-A2 will lead to the unbinding of IGF-1 from its binding proteins and that they will be able to measure free IGF-1 in the blood of this female adult.

DETAILED DESCRIPTION:
PAPP-A2 is a plasma protease that is known to cleave IGFBP-3 and IGFBP-5. It is thought that this cleavage frees up IGF-1 from its bound form allowing it to become the active free IGF-1. The participant has short stature accompanied with elevated plasma levels of both IGF-1 and IGF binding protein 3 (IGFBP-3). Genetic analysis of the participant identified a novel missense mutation in PAPPA2 (Ala1033Val). This gene is a perfect candidate to explain our patients' phenotype. The investigators' hypothesis is that loss of activity of PAPP-A2 leads to an inability to cleave the IGF binding proteins and thus an overall elevation in IGFBP-3 and consequent elevation in total IGF-1. However, this IGF-1 cannot be freed up and is thus not able to be active leading to short stature. The patient's missense variant is predicted to be damaging by in silicon prediction models such as Polyphen2. Furthermore, two knock out mouse models of PAPPA2 as well as a zebrafish knock out exist, all showing growth retardation (post-natally in the mice). Taken together, this is definitive evidence that the patients' mutation in PAPPA2 is responsible for their short stature phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for a defect in PAPPA2.

Exclusion Criteria: None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Decrease in IGF-1 | 5 minutes
  Decrease in either total IGF-1 or IGFBP-3 of 20% or greater as a clinically meaningful decrease in levels

SECONDARY OUTCOMES:
Length of decrease in IGF-1 | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dauber, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States